CLINICAL TRIAL: NCT01698112
Title: Does Flaxseed Supplementation Improve Glycemic Control in Individuals With Pre-diabetes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Andrea Hutchins, Associate Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PreDiabetes Flax; 7-06-RA-61 (Other Grant/Funding Number: American Diabetes Association/7-06-RA-61)
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flaxseed High Dose (Experimental)
  Interventions: Dietary Supplement: Flaxseed High Dose
- Flaxseed Low Dose (Experimental)
  Interventions: Dietary Supplement: Flaxseed Low Dose
- Flaxseed control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Flaxseed High Dose — 26 gram flaxseed intervention
  Arms: Flaxseed High Dose
Dietary Supplement: Flaxseed Low Dose — 13 grams flaxseed
  Arms: Flaxseed Low Dose

SUMMARY:
This project is a clinical intervention trial that will determine the role of a functional food, flaxseed, on the control of blood glucose levels in people with pre-diabetes. People with pre-diabetes have high blood glucose levels since their cells do not respond to insulin as they should. Over time, people with pre-diabetes may progress to type 2 diabetes and have increased risk for heart and kidney diseases. Although the long-term complications associated with type 2 diabetes are well-recognized, clinicians and researchers are now realizing that some long-term damage to the body, especially the heart and circulatory system, may already be occurring during pre-diabetes. Consequently, clinicians are recognizing that glucose control, through diet, exercise and, if necessary, medications, is as important for people with pre-diabetes as it is for people with type 2 diabetes.

Standard treatments for pre-diabetes are glucose control through diet, exercise, and drugs. A possible treatment that could be added to the standard treatments is intake of flaxseed. Few studies have looked at the effect of flaxseed intake on glucose control and those that have enrolled people with type 2 diabetes. To date, no studies have reported flaxseed's affect on controlling blood glucose in people with pre-diabetes. Therefore, more research is needed to determine if flaxseed is an effective means of controlling glucose levels in people with pre-diabetes.

This study will help determine whether or not eating modest amounts of flaxseed every day will improve blood glucose and insulin levels in overweight or obese men and postmenopausal women with pre-diabetes. It will also show if flaxseed intake will reduce the degree of inflammation they are experiencing.

If flaxseed consumption does help control blood glucose levels in people with pre-diabetes and reduce the degree of inflammation they are experiencing, it may help prevent or delay their progression to type 2 diabetes.

DETAILED DESCRIPTION:
Pre-diabetes is characterized by hyperglycemia due to ineffective insulin or 'insulin resistance'. Over time, people with pre-diabetes may progress to type 2 diabetes and experience complications including cardiovascular and peripheral vascular disease, hyperlipidemia, retinopathy, neuropathy, and/or nephropathy. Conventional interventions for pre-diabetes are glucose control through diet, exercise, and, if necessary, medications. An efficient but still uncommon adjunct intervention is flaxseed supplementation. Since few studies have examined the affect of flaxseed supplementation on type 2 diabetes and to date, no studies have reported flaxseed's influence on glycemic control in individuals with pre-diabetes, additional research is warranted. The objective of this study is to determine the affect of consuming flaxseed on fasting plasma glucose, insulin, fructosamine, adiponectin, fatty acid concentrations, serum interleukin-6 (hs-IL-6), C-reactive protein (hs-CRP), and urinary lignan excretion in overweight or obese men and postmenopausal women with pre-diabetes. This research will provide data for the strength of the relationship between regular flaxseed intake and biomarkers for pre-diabetes and glycemic control as well as adiponectin values and markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* (1) no unresolved health conditions (e.g. if high blood pressure is present it is under control due to diet and/or medications) and no diagnosis of type 2 diabetes;
* (2) non-smoking status;
* (3) no regular history of flaxseed or flaxseed oil supplement or fish oil supplement intake;
* (4) no regular history of sunflower seed intake (1/8 cup < 1 time per week); fish intake (< 12 ounces of fish/week); and soy intake (1 serving of soy < 3 times per week; 1 serving of soy equals 3 oz. tofu, 8 oz. soy milk, ¼ c. soy nuts or ½ c. edamame);
* (5) willingness to follow study protocol, scheduling, and testing location;
* (6) body mass index (BMI) of 25-34.9 kg/m2;
* (7) men or postmenopausal women (no menstrual cycle for > 6 months; women who have had a hysterectomy are eligible for participation) ages 50-65 years;
* (8) fasting glucose value of > 100 and < 126 mg/dL.

Exclusion Criteria:

* (1) unresolved health conditions or diagnosis of type 2 diabetes;
* (2) smokes;
* (3) regular history of flaxseed or flaxseed oil supplement or fish oil supplement intake;
* (4) regular history of sunflower seed intake (1/8 cup < 1 time per week); fish intake (< 12 ounces of fish/week); and soy intake (1 serving of soy < 3 times per week; 1 serving of soy equals 3 oz. tofu, 8 oz. soy milk, ¼ c. soy nuts or ½ c. edamame);
* (5) unwillingness to follow study protocol, scheduling, and testing location;
* (6) body mass index (BMI) less than 25 or greater than 34.9 kg/m2;
* (7) premenopausal women;
* (8) men or postmenopausal women less than 50 or greater than 65 years of age;
* (9) fasting glucose value of less than 100 or greater than 126 mg/dL.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | beginning and end of each 12-week intervention (start of 1st week and end of 12th week)
Fasting insulin | beginning and end of each 12-week intervention (start of 1st week and end of 12th week)
Fasting fructosamine | beginning and end of each 12-week intervention (start of 1st week and end of 12th week)

SECONDARY OUTCOMES:
C-reactive protein | beginning and end of each 12-week intervention (start of 1st week and end of 12th week)
interleukin 6 | beginning and end of each 12-week intervention (start of 1st week and end of 12th week)
adiponectin | beginning and end of each 12-week intervention (start of 1st week and end of 12th week)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hutchins, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (2):
- United States (2):
  - University of Colorado Colorado Springs, Colorado Springs, Colorado
  - University of Montana, Missoula, Montana